CLINICAL TRIAL: NCT01667549
Title: Sensitive Periods in Human Flavor Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monell Chemical Senses Center (Other)
Responsible Party: Principal Investigator, Julie A. Mennella, PhD, Member and Director Emeritus, Monell Chemical Senses Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: HD37119
Record Dates: First submitted 2012-08-13; First posted 2012-08-17 (Estimated); Results first posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-11

CONDITIONS: Development
Keywords: Breastfeeding; Flavor learning; Mother; Moms; Infants; Babies; Baby; Food Habits; Fruits; Vegetables
MeSH Terms: conditions — Breast Feeding; Feeding Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1M0.5 (Experimental): Mothers will receive the intervention for 1 month beginning when their infant is 0.5 months old.
  Intervention: Timing of Diet and Flavor Experience
  Interventions: Other: Timing of Diet and Flavor Experience
- 1M1.5 (Experimental): Mothers will receive the intervention for 1 month beginning when their infant is 1.5 months old.
  Intervention: Timing of Diet and Flavor Experience
  Interventions: Other: Timing of Diet and Flavor Experience
- 3M0.5 (Experimental): Mothers will receive the intervention for 3 months beginning when their infant is 0.5 months old.
  Intervention: Timing of Diet and Flavor Experience
  Interventions: Other: Timing of Diet and Flavor Experience
- Control (No Intervention): Mothers will not receive the intervention.

INTERVENTIONS:
Other: Timing of Diet and Flavor Experience — Groups differ in the timing and duration of exposure to flavored food experience.
  Arms: 1M0.5; 1M1.5; 3M0.5

SUMMARY:
The goals of the proposed research are to specify the timing and consequences of the sensitive period for flavor learning in infants who are being breastfed or formula fed. The investigators will conduct a randomized within- and between-subject study of women and their infants during a 15-month window.

DETAILED DESCRIPTION:
This is a randomized clinical trial on both breastfeeding and formula feeding infants to determine the effects of the timing of flavor experiences on subsequent food acceptance in both members of the dyad.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, term infants and their mothers
* Infants 2 wks (+/- 2 wk of age)
* Mothers and infants exclusively breastfeeding or exclusively feeding a cows-milk based formula
* Mothers must be older than 18 years of age

Exclusion Criteria:

* Infants who were preterm or have medical conditions that interfere with feeding or eating
* Mothers who had gestational diabetes or are diagnosed with a major illness requiring treatment or surgery
* Mothers who will be going back to work full-time before the infant is 4 months old
* Mothers who are allergic to any vegetables
* Subjects will not be excluded because of economic status, gender, race or ethnicity.

Ages: 2 Weeks to 3 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 97 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Mennella, PhD, Principal Investigator — Monell Chemical Senses Center
Locations (1):
- Monell Chemical Senses Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available

REFERENCES:
- [Background] Mennella JA, Jagnow CP, Beauchamp GK. Prenatal and postnatal flavor learning by human infants. Pediatrics. 2001 Jun;107(6):E88. doi: 10.1542/peds.107.6.e88. PMID 11389286
- [Background] Skinner JD, Carruth BR, Wendy B, Ziegler PJ. Children's food preferences: a longitudinal analysis. J Am Diet Assoc. 2002 Nov;102(11):1638-47. doi: 10.1016/s0002-8223(02)90349-4. PMID 12449287
- [Background] Mennella JA, Lukasewycz LD, Castor SM, Beauchamp GK. The timing and duration of a sensitive period in human flavor learning: a randomized trial. Am J Clin Nutr. 2011 May;93(5):1019-24. doi: 10.3945/ajcn.110.003541. Epub 2011 Feb 10. PMID 21310829
- [Background] Mennella JA, Pepino MY, Reed DR. Genetic and environmental determinants of bitter perception and sweet preferences. Pediatrics. 2005 Feb;115(2):e216-22. doi: 10.1542/peds.2004-1582. PMID 15687429
- [Background] Forestell CA, Mennella JA. Early determinants of fruit and vegetable acceptance. Pediatrics. 2007 Dec;120(6):1247-54. doi: 10.1542/peds.2007-0858. PMID 18055673
- [Background] Llewellyn CH, van Jaarsveld CH, Johnson L, Carnell S, Wardle J. Development and factor structure of the Baby Eating Behaviour Questionnaire in the Gemini birth cohort. Appetite. 2011 Oct;57(2):388-96. doi: 10.1016/j.appet.2011.05.324. Epub 2011 Jun 6. PMID 21672566
- [Background] Pliner P, Hobden K. Development of a scale to measure the trait of food neophobia in humans. Appetite. 1992 Oct;19(2):105-20. doi: 10.1016/0195-6663(92)90014-w. PMID 1489209
- [Background] Gerrish CJ, Mennella JA. Flavor variety enhances food acceptance in formula-fed infants. Am J Clin Nutr. 2001 Jun;73(6):1080-5. doi: 10.1093/ajcn/73.6.1080. PMID 11382663
- [Background] Mennella JA, Nicklaus S, Jagolino AL, Yourshaw LM. Variety is the spice of life: strategies for promoting fruit and vegetable acceptance during infancy. Physiol Behav. 2008 Apr 22;94(1):29-38. doi: 10.1016/j.physbeh.2007.11.014. Epub 2007 Nov 21. PMID 18222499
- [Derived] Mennella JA, Reiter A, Brewer B, Pohlig RT, Stallings VA, Trabulsi JC. Early Weight Gain Forecasts Accelerated Eruption of Deciduous Teeth and Later Overweight Status during the First Year. J Pediatr. 2020 Oct;225:174-181.e2. doi: 10.1016/j.jpeds.2020.06.019. Epub 2020 Jun 15. PMID 32553836
- [Derived] Mennella JA, Daniels LM, Reiter AR. Learning to like vegetables during breastfeeding: a randomized clinical trial of lactating mothers and infants. Am J Clin Nutr. 2017 Jul;106(1):67-76. doi: 10.3945/ajcn.116.143982. Epub 2017 May 17. PMID 28515063

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pregnant women or newly parturient women who intended to breastfeed their infants exclusively for at least 4 months were recruited from ads in local newspapers, websites, and Philadelphia Women, Infants, and Children (WIC) offices. We enroll mother -infant dyads because both members of the dyads were tested.
Pre-assignment Details: No mother-infant dyads were excluded from the study prior to assignment to groups.
Groups:
- 1M0.5: Mothers will receive the intervention for 1 month beginning when their infant is 0.5 months old.
  Intervention: Timing of Diet and Flavor Experience
  Timing of Diet and Flavor Experience: Groups differ in the timing and duration of exposure to flavored food experience.
- 1M1.5: Mothers will receive the intervention for 1 month beginning when their infant is 1.5 months old.
  Intervention: Timing of Diet and Flavor Experience
  Timing of Diet and Flavor Experience: Groups differ in the timing and duration of exposure to flavored food experience.
- 1M2.5: Mothers will receive the intervention for one month beginning when their infants are 2.5 months of age
- 3M0.5: Mothers will receive the intervention for 3 months beginning when their infant is 0.5 months old.
  Intervention: Timing of Diet and Flavor Experience
  Timing of Diet and Flavor Experience: Groups differ in the timing and duration of exposure to flavored food experience.
Period: Overall Study
Arm/Group | 1M0.5 | 1M1.5 | 1M2.5 | 3M0.5 | Control
Started | 20 (20 dyads=20 infants, 20 mothers) | 20 (20 dyads=20 infants, 20 mothers) | 21 (21 dyads=21 infants, 21 mothers) | 20 (20 dyads= 20 infants, 20 mothers) | 16 (16 dyads=16 infants, 16 mothers)
Completed | 17 (17 dyads=17 infants, 17 mothers) | 15 (15 dyads=15 infants, 15 mothers) | 14 (14 dyads=14 infants, 14 mothers) | 14 (14 dyads= 14 infants, 14 mothers) | 15 (15 dyads=15 infants, 15 mothers)
Not Completed | 3 | 5 | 7 | 6 | 1
Not completed — Withdrawal by Subject | 3 | 5 | 7 | 6 | 1

BASELINE CHARACTERISTICS:
Population: The number of baseline participants refers to number of infants or number of mothers, depending on outcome
Groups:
- 1M2.5: Mothers will receive the intervention for one month beginning when their infants are 2.5 months old.
  Intervention: Timing of Diet and Flavor Experience
  Timing of Diet and Flavor Experience: Groups differ in the timing and duration of exposure to flavored food experience.
- Total: Total of all reporting groups
Arm/Group | 1M0.5 | 1M1.5 | 1M2.5 | 3M0.5 | Control | Total
Number analyzed (Participants) | 20 | 20 | 21 | 20 | 16 | 97
Age, Continuous [Mean (Standard Deviation); unit: Months] — Population: Dyads consists of mothers and their infants and different measures were obtained from each.
  Months
    Infants' Age in months | 0.5 (0.1) | 0.6 (0.1) | 0.6 (0.1) | 0.6 (0.1) | 0.5 (0.1) | 0.5 (0.1)
Age, Continuous [Mean (Standard Deviation); unit: Mothers' Age in years] | 32.5 (4.4) | 30.5 (6.2) | 29.8 (5.2) | 29.9 (5.1) | 31.7 (5.9) | 30.8 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants] — The genotype of infants are reported separately from mothers. Genotyping was attempted but failed for one infant. Population: Infants are reported separately from mothers
  Participants
    Sex of Infants: Female | 10 | 11 | 9 | 13 | 7 | 50
    Sex of Infants: Male | 10 | 9 | 12 | 7 | 9 | 47
    Sex of Mothers: Female | 20 | 20 | 21 | 20 | 16 | 97
    Sex of Mothers: Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Infants are reported separately from mothers.
  Participants
    Infants: Hispanic or Latino | 2 | 4 | 4 | 3 | 1 | 14
    Infants: Not Hispanic or Latino | 18 | 16 | 17 | 17 | 15 | 83
    Infants: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
    Mothers: Hispanic or Latino | 2 | 3 | 2 | 2 | 0 | 9
    Mothers: Not Hispanic or Latino | 18 | 17 | 19 | 18 | 16 | 88
    Mothers: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Infants are reported separately from mothers.
  Participants
    Infants: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
    Infants: Asian | 0 | 1 | 0 | 0 | 1 | 2
    Infants: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
    Infants: Black or African American | 3 | 7 | 8 | 8 | 5 | 31
    Infants: White | 13 | 9 | 9 | 9 | 9 | 49
    Infants: More than one race | 4 | 3 | 4 | 3 | 1 | 15
    Infants: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
    Mothers: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
    Mothers: Asian | 0 | 1 | 0 | 0 | 1 | 2
    Mothers: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
    Mothers: Black or African American | 4 | 7 | 10 | 9 | 5 | 35
    Mothers: White | 14 | 9 | 11 | 10 | 10 | 54
    Mothers: More than one race | 2 | 3 | 0 | 1 | 0 | 6
    Mothers: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Genotype, TAS2R38 taste gene [secondary outcome] [Count of Participants; unit: Participants] — Population: Infants are reported separately from their mothers. Genotyping was unsuccessful for one infant.
  Participants
    Infants: TAS2R38 genotype, AA [non taster] | 7 | 6 | 3 | 7 | 8 | 31
    Infants: TAS2R38 genotype AP [taster, heterozygote] | 12 | 8 | 11 | 7 | 5 | 43
    Infants: TAS2R38 genotype PP [taster] | 1 | 6 | 7 | 6 | 2 | 22
    Infants: Genotyping unsuccessful | 0 | 0 | 0 | 0 | 1 | 1
    Mothers: TAS2R38 genotype, AA [non taster] | 4 | 5 | 5 | 7 | 11 | 32
    Mothers: TAS2R38 genotype AP [taster, heterozygote] | 12 | 9 | 9 | 8 | 3 | 41
    Mothers: TAS2R38 genotype PP [taster] | 4 | 6 | 7 | 5 | 2 | 24
    Mothers: Genotyping unsuccessful | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Vegetable Flavor Acceptance [Infants' Intake]
Description: Taste testing conducted on infants to determine acceptance of plain cereal, carrot-flavor cereal (exposed flavor for intervention groups) and broccoli-flavored cereal (novel flavor for all groups) after weaning, which occurred at ~ 8 months of age. Outcomes included intake (in grams).
Time Frame: 6- to 10-month-old weaned infants (3 separate test days )
Population: Some of the infants refused to eat (plain cereal: 1M0.5, N=1; 1M1.5, N=1; 1M2.5, N=4; 3M0.5, N=1; carrot cereal: 1M0.5, N=2; 1M1.5, N=2; 1M2.5, N=4; 3M0.5, N=1; Broccoli: 1M0.5, N=1; 1M1.5, N=1; 1M2.5, N=3; 3M0.5 , N=1) and therefore the number participants analyzed differs from number in each group
Measure: Mean (Standard Error); unit: intake in grams
Arm/Group | 1M0.5 | 1M1.5 | 1M2.5 | 3M0.5 | Control
Number analyzed (Participants) | 17 | 15 | 14 | 14 | 15
intake in grams
  Intake of plain cereal in grams: number analyzed (Participants) | 16 | 14 | 10 | 13 | 15
  Intake of plain cereal in grams | 56.8 (13.2) | 42.4 (12.4) | 29.0 (8.5) | 40.7 (8.3) | 36.5 (6.2)
  Intake of carrot cereal in grams: number analyzed (Participants) | 15 | 13 | 10 | 13 | 15
  Intake of carrot cereal in grams | 78.2 (14.8) | 36.6 (10.0) | 57.7 (19.9) | 52.2 (9.8) | 41.1 (7.6)
  Intake of broccoli cereal, grams: number analyzed (Participants) | 16 | 14 | 11 | 13 | 15
  Intake of broccoli cereal, grams | 41.8 (12.7) | 25.5 (8.8) | 30.9 (10.1) | 34.4 (12.4) | 3.04 (6.5)
Statistical Analysis 1: Comparison: 1M0.5 vs 1M1.5 vs 1M2.5 vs 3M0.5; Separate analyses of variance with a priori contrasts specified were conducted: 1) to determine whether the 1-month exposure groups (1M0.5, 1M1.5, and 1M2.5) differed from the no-exposure control group to test the hypothesis that the timing of exposure affected acceptance; and 2) to determine whether 1 month of exposure differed from 3 months (1M0.5, 3M0.5 groups) and whether these groups differed from the no-exposure control group (duration hypothesis); Test type: Other — Repeated Measures ANOVA were done with type of cereal as within-subjects and experimental group as grouping factors. When significant, planned comparisons were carried out. ANOVAs with a priori contrasts specified determined whether 1-month exposure differed from the no-exposure control (timing hypothesis). ANOVAs with a priori contrasts specified determined whether 1-month differed from 3-months exposure and whether these groups differed from no-exposure control (duration hypothesis); p = 0.02, planned comparison — Bonferroni adjustment was made and only planned pairwise comparisons with calculated p values of 0.02 or lower significant; Bonferroni adjustment was calculated and only planned pair-wise comparisons with calculated p value 0.02 or lower were considered significant

2. Primary Outcome: Taste Liking Ratings of Vegetable Flavors [Mothers].
Description: Psychophysical testing conducted on mothers to rate their taste of carrot, beet, celery, mixed vegetable (exposed flavors for intervention groups) and apple juices using the hedonic gLMS (hedonic general labelled magnitude scale). Ratings on the scale range from -100 (strongest imaginable dislike) to 0 (neutral) to 100 (strongest imaginable like).
Time Frame: Monthly, 0.5 to 4.5 months
Population: Two mothers did not complete the ratings on one test date.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | 1M0.5 | 1M1.5 | 1M2.5 | 3M0.5 | Control
Number analyzed (Participants) | 17 | 15 | 14 | 14 | 15
units on a scale
  Carrot, 0.5 mos (baseline) | -0.07 (4.84) | -3.35 (5.15) | -1.28 (5.33) | -2.02 (5.33) | -4.71 (5.15)
  Carrot, 1.5 mos | 6.21 (3.41) | 1.28 (3.63) | 3.91 (3.75) | 4.17 (3.75) | 1.46 (3.63)
  Carrot, 2.5 mos | 5.67 (3.19) | 3.51 (3.39) | 2.08 (3.51) | 6.30 (3.51) | -2.53 (3.39)
  Carrot, 3.5 mos: number analyzed (Participants) | 17 | 14 | 14 | 14 | 15
  Carrot, 3.5 mos | 3.10 (3.36) | 6.20 (3.71) | 7.78 (3.7) | 3.05 (3.71) | 1.56 (3.58)
  Carrot, 4.5 mos: number analyzed (Participants) | 17 | 14 | 14 | 14 | 15
  Carrot, 4.5 mos | 5.86 (3.35) | 4.82 (3.69) | 6.20 (3.69) | 2.63 (3.69) | 2.75 (3.57)
  Beet, 0.5 mos (baseline) | 5.81 (5.37) | 1.18 (5.72) | -0.65 (5.92) | 0.87 (5.92) | -3.21 (5.72)
  Beet, 1.5 mos | 3.13 (4.16) | 9.35 (4.43) | -2.20 (4.58) | 3.40 (4.58) | 5.73 (4.43)
  Beet, 2.5 mos | 9.29 (3.50) | 6.41 (3.73) | -0.68 (3.86) | 1.02 (3.86) | 9.17 (3.73)
  Beet, 3.5 mos: number analyzed (Participants) | 17 | 14 | 14 | 14 | 15
  Beet, 3.5 mos | 10.87 (3.94) | 7.74 (4.34) | 7.54 (4.34) | 3.52 (4.34) | 6.82 (4.20)
  Beet, 4.5 mos: number analyzed (Participants) | 17 | 14 | 14 | 14 | 15
  Beet, 4.5 mos | 8.63 (3.48) | 10.34 (3.83) | 9.35 (3.83) | 3.58 (3.83) | 7.89 (3.70)
  Mixed Vegetables, 0.5 mos (baseline) | 1.22 (5.05) | 0.20 (5.38) | 0.82 (5.57) | 0.97 (5.57) | 11.32 (5.38)
  Mixed Vegetables, 1.5 mos | 9.48 (3.96) | 0.18 (4.22) | 1.11 (4.36) | 4.30 (4.36) | 10.69 (4.22)
  Mixed Vegetables, 2.5 mos | 10.19 (3.31) | 6.32 (3.52) | 2.23 (3.65) | 6.14 (3.65) | 7.57 (3.52)
  Mixed Vegetables, 3.5 mos: number analyzed (Participants) | 17 | 14 | 14 | 14 | 15
  Mixed Vegetables, 3.5 mos | 7.00 (3.52) | 5.69 (3.88) | 3.81 (3.88) | 6.01 (3.88) | 10.42 (3.75)
  Mixed Vegetables, 4.5 mos: number analyzed (Participants) | 17 | 14 | 14 | 14 | 15
  Mixed Vegetables, 4.5 mos | 8.40 (3.32) | 6.83 (3.66) | 1.02 (3.66) | 3.62 (3.66) | 7.87 (3.54)
  Celery, 0.5 mos (baseline) | 0.59 (4.72) | -5.33 (5.02) | -13.35 (5.20) | -12.46 (5.20) | -10.36 (5.02)
  Celery, 1.5 mos | -3.93 (3.86) | -0.90 (3.92) | -13.48 (4.06) | -9.68 (4.06) | -5.44 (3.92)
  Celery, 2.5 mos | -0.92 (3.99) | -0.51 (4.24) | -3.01 (4.39) | -6.20 (4.39) | -2.88 (4.24)
  Celery, 3.5 mos: number analyzed (Participants) | 17 | 14 | 14 | 14 | 15
  Celery, 3.5 mos | -5.12 (3.72) | 1.07 (4.10) | -10.40 (4.10) | -8.07 (4.10) | -6.69 (3.96)
  Celery, 4.5 mos: number analyzed (Participants) | 17 | 14 | 14 | 14 | 15
  Celery, 4.5 mos | -6.15 (3.77) | -1.44 (4.16) | -5.89 (4.16) | -5.87 (4.16) | -2.91 (4.02)
  Apple, 0.5 mos (Baseline) | 17.85 (3.64) | 17.48 (3.88) | 22.41 (4.02) | 14.57 (4.02) | 23.72 (3.88)
  Apple, 1.5 mos | 17.04 (2.98) | 20.08 (3.17) | 11.81 (3.28) | 18.23 (3.28) | 20.36 (3.17)
  Apple, 2.5 months | 18.09 (2.95) | 15.97 (3.15) | 17.91 (3.26) | 16.72 (3.26) | 19.39 (3.15)
  Apple, 3.5 mos: number analyzed (Participants) | 17 | 14 | 14 | 14 | 15
  Apple, 3.5 mos | 13.39 (3.52) | 22.56 (3.88) | 17.01 (3.88) | 19.56 (3.88) | 19.44 (3.75)
  Apple, 4.5 months: number analyzed (Participants) | 17 | 14 | 14 | 14 | 15
  Apple, 4.5 months | 15.89 (2.73) | 19.87 (3.01) | 15.45 (3.01) | 19.94 (3.01) | 22.06 (2.91)
Statistical Analysis 1: Comparison: 1M0.5 vs 1M1.5 vs 1M2.5 vs 3M0.5; Repeated measures ANOVAs were conducted on maternal gLMS ratings with type of juice and time as the within-subject factors and experimental group as the grouping factor; Test type: Other; p < 0.02, ANOVA

3. Primary Outcome: Vegetable Flavor Acceptance (Infants' Rate of Feeding)
Description: Taste testing conducted on infants to determine acceptance of plain cereal, carrot-flavor cereal (exposed flavor for intervention groups) and broccoli-flavored cereal (novel flavor for all groups) after weaning, which occurred at ~ 8 months of age. Outcomes included intake rate of feeding (grams per minute) .
Time Frame: 6- to 10-month-old weaned infants (3 separate test days)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: grams per minute
Groups:
- 1M0.5: Mothers received the intervention for 1 month beginning when their infant was 0.5 months old.
  Intervention: Timing of Diet and Flavor Experience
  Timing of Diet and Flavor Experience: Groups differ in the timing and duration of exposure to flavored food experience.
- 1M1.5: Mothers received the intervention for 1 month beginning when their infant was 1.5 months old.
  Intervention: Timing of Diet and Flavor Experience
  Timing of Diet and Flavor Experience: Groups differ in the timing and duration of exposure to flavored food experience.
- 1M2.5: Mothers received the intervention for 1 month beginning when their infant was 2.5 months old.
  Intervention: Timing of Diet and Flavor Experience
  Timing of Diet and Flavor Experience: Groups differ in the timing and duration of exposure to flavored food experience.
- 3M0.5: Mothers received the intervention for 3 months beginning when their infant was 0.5 months old.
  Intervention: Timing of Diet and Flavor Experience
  Timing of Diet and Flavor Experience: Groups differ in the timing and duration of exposure to flavored food experience.
- Control: Mothers did not receive the intervention.
Arm/Group | 1M0.5 | 1M1.5 | 1M2.5 | 3M0.5 | Control
Number analyzed (Participants) | 17 | 15 | 14 | 14 | 15
grams per minute
  Rate of feeding, plain cereal: number analyzed (Participants) | 16 | 14 | 10 | 13 | 15
  Rate of feeding, plain cereal | 6.1 (0.9) | 3.9 (1.1) | 4.0 (0.8) | 4.3 (0.4) | 4.9 (0.6)
  Rate of feeding, carrot cereal: number analyzed (Participants) | 15 | 13 | 10 | 13 | 15
  Rate of feeding, carrot cereal | 7.2 (1.1) | 3.6 (0.8) | 4.8 (1.3) | 3.9 (0.5) | 3.9 (0.6)
  Rate of feeding, broccoli cereal: number analyzed (Participants) | 16 | 14 | 11 | 13 | 15
  Rate of feeding, broccoli cereal | 4.8 (0.8) | 2.4 (0.9) | 4.5 (1.0) | 3.8 (0.9) | 4.1 (0.8)
Statistical Analysis 1: Comparison: 1M0.5 vs 1M1.5 vs 1M2.5 vs 3M0.5; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.02, planned comparison — Because three comparisons were made for each outcome measure, a Bonferroni adjustment was calculated and only planned comparison with P's<0.02 were considered significant; a Bonferroni adjustment was calculated and only planned comparison with P's<0.02 were considered significant

4. Secondary Outcome: Maternal Perceptions
Description: Mothers rated infants' enjoyment of the taste of the cereal (9-point scale); aratings range from 1 (extreme dislike) to 9 (extreme like).
Time Frame: 6- to 10-month-old weaned infants (3 separate test days)
Population: Some of the infants refused to eat (plain cereal: 1M0.5, N=1; 1M1.5, N=1; 1M2.5, N=4; 3M0.5, N=1; carrot cereal: 1M0.5, N=2; 1M1.5, N=2; 1M2.5, N=4; 3M0.5, N=1; Broccoli: 1M0.5, N=1; 1M1.5, N=1; 1M2.5, N=3; 3M0.5 , N=1) and therefore the number of maternal ratings analyzed differs from number in each group
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | 1M0.5 | 1M1.5 | 1M2.5 | 3M0.5 | Control
Number analyzed (Participants) | 17 | 15 | 14 | 14 | 15
Score on a scale
  Rating of infant enjoyment, plain cerea: number analyzed (Participants) | 16 | 14 | 10 | 13 | 15
  Rating of infant enjoyment, plain cerea | 5.4 (0.6) | 4.6 (0.8) | 4.1 (0.9) | 5.2 (0.6) | 3.9 (0.5)
  Rating of infant enjoyment, carrot cereal: number analyzed (Participants) | 15 | 13 | 10 | 13 | 15
  Rating of infant enjoyment, carrot cereal | 6.0 (0.7) | 4.7 (0.7) | 7.1 (0.4) | 6.1 (0.5) | 6.1 (0.7)
  Rating of infant enjoyment, broccoli cere: number analyzed (Participants) | 16 | 14 | 11 | 13 | 15
  Rating of infant enjoyment, broccoli cere | 4.2 (0.7) | 2.9 (0.6) | 4.7 (0.7) | 4.3 (0.6) | 4.1 (0.7)
Statistical Analysis 1: Comparison: 1M0.5 vs 1M1.5 vs 1M2.5 vs 3M0.5 vs Control; Separate analyses of variance with a priori contrasts specified 1) to determine whether the 1-month exposure groups (1M0.5, 1M1.5, and 1M2.5) differed from the no-exposure control group to test the hypothesis that the timing of exposure affected acceptance; and 2) to determine whether 1 month of exposure differed from 3 months (1M0.5, 3M0.5 groups) and whether these groups differed from the no-exposure control group (duration hypothesis); Test type: Other; p < 0.02, planned comparison — Because three comparisons were made for each outcome measure, a Bonferroni adjustment was calculated and only planned comparison with P<0.02 were considered significant; A Bonferroni adjustment was calculated and only planned comparison with P's<0.02 were considered significant

5. Secondary Outcome: Growth of Infants
Description: At each visit, infants were weighed and measured to monitor normal growth. These anthropometric data were converted to weight-for-length z-scores (WLZ) using World Health Organization (WHO) growth standards. The Z-score expresses the anthropometric value as a number of standard deviations or Z-scores below or above the reference mean or median value. Normal range for Z score is -2.0 (minimum) to 2.0 (maximum).
Time Frame: Once a month from ages 0.5 - 4.5 months, 10.5 months
Population: Number of infants who were weighted and measured to determine Weight for Length Z scores (WLZ) during trial; some dyads did not complete the trial so number of participants analyzed does not always match number enrolled.
Measure: Mean (Standard Error); unit: Z score
Arm/Group | 1M0.5 | 1M1.5 | 1M2.5 | 3M0.5 | Control
Number analyzed (Participants) | 17 | 15 | 14 | 14 | 15
Z score
  Weight for Length Z: 0.5 months | -0.69 (0.24) | 0.04 (0.26) | -0.40 (0.27) | 0.10 (0.27) | -0.56 (0.26)
  Weight for Length Z: 1.5 months | -0.07 (0.27) | 0.42 (0.28) | -0.49 (0.29) | 0.56 (0.29) | 0.14 (0.28)
  Weight for Length Z: 2.5 months: number analyzed (Participants) | 17 | 14 | 14 | 14 | 15
  Weight for Length Z: 2.5 months | 0.04 (0.26) | 0.13 (0.29) | -0.64 (0.29) | 0.45 (0.29) | 0.15 (0.28)
  Weight for Length Z: 3.5 months: number analyzed (Participants) | 17 | 14 | 14 | 14 | 15
  Weight for Length Z: 3.5 months | 0.02 (0.28) | 0.12 (0.31) | -0.68 (0.31) | 0.63 (0.31) | 0.08 (0.30)
  Weight for Length Z: 4.5 months: number analyzed (Participants) | 17 | 14 | 14 | 14 | 14
  Weight for Length Z: 4.5 months | 0.20 (0.25) | 0.05 (0.27) | -0.67 (0.27) | 0.43 (0.27) | 0.30 (0.27)
  Weight for Length Z, 10.5 months: number analyzed (Participants) | 17 | 14 | 14 | 14 | 15
  Weight for Length Z, 10.5 months | 0.56 (0.24) | 0.67 (0.26) | 0.23 (0.26) | 0.61 (0.26) | 0.54 (0.25)
Statistical Analysis 1: Comparison: 1M0.5 vs 1M1.5 vs 1M2.5 vs 3M0.5 vs Control; General linear models were conducted on WLZ scores with time as the within-subjects factor and Group as the between-subjects factor to determine there were differences in growth of the infants over time. This was not done to test hypothesis but to monitor growth of infants during course of trial; Test type: Other; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | 1M0.5 | 1M1.5 | 1M2.5 | 3M0.5 | Control
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/21 | 0/20 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/21 | 0/20 | 0/16
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/21 | 0/20 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No